CLINICAL TRIAL: NCT05117294
Title: A Phase 1 Open Label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ASP0367 in Participants With Renal Impairment Compared to Healthy Participants With Normal Renal Function
Brief Title: A Study of ASP0367 in People With Kidneys That do Not Work Well and in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0367-CL-1111; 2021-004042-38 (EudraCT Number)
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Renal Impairment; Healthy Volunteers
Keywords: Severe renal impairment; Moderate renal impairment; Mild renal impairment; ASP0367; Pharmacokinetics; Healthy Volunteers; MA-0211; Kidney function; Bocidelpar
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bocidelpar (ASP0367): Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single dose of Bocidelpar (ASP0367) under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar
- Bocidelpar (ASP0367): Moderate Renal Impairment (Experimental): Participants with moderate renal impairment will receive a single dose of Bocidelpar (ASP0367) under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar
- Bocidelpar (ASP0367): Mild Renal Impairment (Experimental): Participants with mild renal impairment will receive a single dose of Bocidelpar (ASP0367) under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar
- Bocidelpar (ASP0367): Normal Renal Function (Experimental): Participants with normal renal function will receive a single dose of Bocidelpar (ASP0367) under fasting conditions on day 1.
  Interventions: Drug: Bocidelpar

INTERVENTIONS:
Drug: Bocidelpar — Oral
  Other Names: MA-0211, ASP0367

SUMMARY:
This study is for adults whose kidneys do not work well (renal impairment) and adults whose kidneys work normally. This study will provide more information on a potential new treatment, called ASP0367. The main aim of the study is to learn how ASP0367 is processed by the body in these different groups of people.

This study will be in 2 parts. Part 2 will only happen if the results between the 2 groups are different in Part 1. In each part, people in the study will stay in a research unit for 6 days and 5 nights. Later, they will return to the research unit for 1 check-up.

In Part 1, people whose kidneys work normally and people whose kidneys work very poorly (severe renal impairment) can take part.

If Part 2 happens, people whose kidneys work normally and people whose kidneys do not work well (mild or moderate renal impairment) can take part.

In both parts of the study, people who can take part will be admitted to the research unit. The next day they will take tablets of ASP0367 just once. People will give blood and urine samples at various times during their stay. They will have their vital signs (heart rate and blood pressure) checked regularly. People will also have ECGs to check their heart rhythm. They will be asked if they have any medical problems. After 6 days, provided all the checks have been done and there are no medical problems, people in the study will leave the research unit.

People will return to the research unit for 1 check-up. This will be between 9 and 11 days after their last blood sample was taken during their previous stay in the unit. The check-up will include a physical exam, a check of people's vital signs (heart rate and blood pressure), and blood tests. Also, people will have an ECG and be asked if they have had any medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index range of 18.5 to 40.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of child-bearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 28 days after Investigational Product (IP) administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 28 days after IP administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 28 days after IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 28 days after IP administration.
* Male participant must not donate sperm during the treatment period and for 28 days after IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 28 days after IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study.
* Participant has normal renal function as defined by estimated glomerular filtration rate (eGFR) using Modification of Diet in Renal Disease formula ≥ 90 mL/min per 1.73 m^2 or participant has varying degrees of chronic kidney disease as defined by the National Kidney Foundation and by eGFR:

  * 60 to < 90 mL/min per 1.73 m^2 for participants with mild renal impairment
  * 30 to < 60 mL/min per 1.73 m^2 for participants with moderate renal impairment
  * < 30 mL/min per 1.73 m^2 and not on hemodialysis, with approximately 50 percent of participants to have eGFR ≤ 20 mL/min per 1.73 m^2 for participants with severe renal impairment
* Participant has adequate venous access.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to day -1.
* Participant has any condition, which makes the participant unsuitable for study participation.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has a known or suspected hypersensitivity to ASP0367 or any components of the formulation used.
* Participant has had previous exposure with ASP0367.
* Participant has used moderate or strong inducers of Cytochrome P450 (CYP) 3A within the 3 months prior to day -1.
* Participant has used a strong CYP3A inhibitor within 5 half lives, prior to day -1.
* Participant has used proton pump inhibitor within the 2 weeks prior to IP administration.
* Participant has used histamine 2 blockers within 24 hours prior to IP administration.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has any of the liver function tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and total bilirubin ≥ 1.5 × upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant is an employee of Astellas, the study related contract research organization (CRO) or the clinical unit.
* Participant has a positive result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction (PCR) test at screening.
* Participant has consumed grapefruit, Seville oranges, grapefruit containing products or Seville orange containing products within 72 hours prior to day -1.
* Participant has a history of smoking > 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1, unless the positive result is due to an approved prescription medication (for participants with renal impairment only).
* For US sites: Participant has a history of consuming > 14 units for male participants or > 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* For EU sites: Participant has a history of consuming > 21 units for male participants or > 14 units for female participants of alcohol per week within 3 months prior to day -1 (note: 1 unit = 10 g pure alcohol, 250 mL of beer [5 percent], 35 mL of spirits [35 percent] or 100 mL of wine [12 percent]) or the participant tests positive for alcohol at screening or on day -1.
* Participant has received a coronavirus disease 2019 (COVID-19) vaccine within the 2 weeks prior to IP administration or will have a COVID-19 vaccine dose before the end-of-study visit (ESV).
* Participant has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.

Participant with renal impairment will be excluded from participation in the study if any of the following apply:

* Participant has a history of any clinically significant illness (other than renal disease and conditions related to the renal disease, such as stable diabetes and stable hypertension), medical condition or laboratory abnormality within 3 months prior to screening.
* Participant has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure (SBP) < 90 or > 160 mmHg; mean diastolic blood pressure (DBP) < 50 or > 100 mmHg (measurements taken in triplicate after participant has been resting in a supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QT interval using Fridericia's correction (QTcF) of > 450 msec (for male participants) and > 480 msec (for female participants) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate may be taken.
* Participant who has had a change in dose regimen of medically required medication(s) in the 2 weeks prior to screening (permitted concomitant medications) and/or participant for whom dose changes are likely to occur during the study (minor dose changes are allowed in agreement with the sponsor) and/or participant has used nonpermitted concomitant medication(s) in the 3 weeks prior to admission to the clinical unit.
* Participant who has a renal disease secondary to malignancy.
* Participant who has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to IP administration, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the screening period.
* Participant has a hemoglobin result of < 9 g/dL.
* Participant has a functioning kidney transplant.
* Participant has cardiac troponin I (cTnI) for a given manufacturer's assay being used that is above the historical upper range for participants with chronic kidney injury in the presence of cardiac symptoms or acute ECG changes suggestive of myocardial infarction or an increase in cTnI by >20% from baseline value at the 2-hour time point at screening.

Healthy participants with normal renal function will be excluded from participation in the study if any of the following apply:

* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean QTcF of > 430 msec (for male participants) and > 450 msec (for female participants) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products), hormonal contraceptives and hormone replacement therapy.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Participant has cardiac troponin (cTnI) > Upper limit of normal (ULN) (or cardiac troponin T [cTnT] > ULN if cTnI is not available) at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of Bocidelpar (ASP0367) in Plasma: Area Under The Concentration-time Curve From Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 5 days
  AUCinf will be recorded from PK plasma samples collected.
Pharmacokinetics (PK) of Bocidelpar (ASP0367) in Plasma: Area Under The Concentration-time Curve From The Time of Dosing to The Last Measurable Concentration (AUClast) | Up to 5 days
  AUClast will be recorded from PK plasma samples collected.
Pharmacokinetics (PK) of Bocidelpar (ASP0367) in Plasma: maximum concentration (Cmax) | Up to 5 days
  Cmax will be recorded from PK plasma samples collected.
Pharmacokinetics (PK) of Bocidelpar (ASP0367) in Plasma: apparent clearance (CL/F) | Up to 5 days
  CL/F will be recorded from PK plasma samples collected.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 16
  Adverse Events (AEs) will be coded using MedDRA. An AE is any untoward medical occurrence in a participant, temporally associated with the use of study IP, whether or not considered related to the study IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants with Laboratory Value Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with Vital Sign Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant vital signs values.
Number of Participants with 12-Lead Electrocardiogram (ECG) Abnormalities and/or AEs | Up to Day 16
  Number of participants with potentially clinically significant 12-Lead ECG values.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (4):
  - Pinnacle Research Group, Anniston, Alabama
  - Inland Empire, Rialto, California
  - Advanced Pharma CR, LLC, Miami, Florida
  - Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.